CLINICAL TRIAL: NCT04222647
Title: Prospective, Open-label, Monocenter, Trial to Investigate the Efficacy and Tolerability of WO533, a Lactic Acid Containing Vaginal Suppository, in a Panel of Post-menopausal Women Suffering From Vulvovaginal Atrophy (VVA)
Brief Title: Investigation of Efficacy and Tolerability of a Lactic Acid Containing Vaginal Suppository in Post-menopausal Women With VVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: proDERM Institut für Angewandte Dermatologische Forschung GmbH (Unknown); Bremer Pharmacovigilance Service GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMP-03/2018; 2019-002325-30 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2020-01-10 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO533 (Experimental): Formulation containing WO533 for intravaginal application
  Interventions: Drug: WO533

INTERVENTIONS:
Drug: WO533 — Intravaginal application

SUMMARY:
The aim of the study is to investigate the efficacy and tolerability of a lactic acid containing vaginal suppository with respect to the application in post-menopausal women with VVA.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with subjective symptomatology of vulvovaginal atrophy
* Signed written informed consent before participation in the trial

Exclusion Criteria:

* Known hypersensitivity against any of the ingredients of the investigational product
* Systemic hormonal replacement therapy, or phytohormonal therapy or use of SERMs within 3 months before and / or during the conduct of the trial
* Local hormonal therapy (vagina/vulva) within 3 months before the trial
* If in the opinion of the investigator the patient should not participate in the study for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
VMI | Day 1 to 43
  Change of the Vaginal Maturation Index (VMI)

SECONDARY OUTCOMES:
Vaginal pH | Day 1 to 8, day 8 to 43, and day 1 to 43
  Change of vaginal pH
Subjective vulvovaginal atrophy symptoms | Day 1 to 8, day 8 to 43, and day 1 to 43
  Change of severity scoring for each of the subjective symptoms (dryness, itching, burning and pain unrelated to sexual intercourse) and as sum score
Global judgment of the tolerability by the Investigator | Day 1 to 43
  Scoring on a scale from 1 to 4
Global judgment of the tolerability by the patient | Day 1 to 43
  Scoring on a scale from 1 to 4
Adverse events | Day 1 to 43

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, MD, Principal Investigator — proDERM Institute for Applied Dermatological Research, Germany
Locations (1):
- proDERM Institute for Applied Dermatological Research, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabes M, Donhauser T, Harder A, Masur C, Apfelbacher CJ. Psychometric evaluation of the German Day-to-Day Impact of Vaginal Aging questionnaire using data from two intervention studies. Menopause. 2023 May 1;30(5):551-555. doi: 10.1097/GME.0000000000002161. Epub 2023 Feb 14. PMID 36787527